CLINICAL TRIAL: NCT03126136
Title: Predictive Value of a Postural Test on Pulse Pressure Variation During Labor With Epidural Analgesia on Fetal Heart Rate Abnormalities
Brief Title: Pulse Pressure Variability With Position Before EPIdural Analgesia
Acronym: PP-PERI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/31; 2016- A00846-45 (Other: ANSM)
Record Dates: First submitted 2017-03-21; First posted 2017-04-24 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Labor; Epidural Analgesia
Keywords: Fetal heart rate abnormalities; Pregnancy; Epidural analgesia; Pulse pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant women (Experimental)
  Interventions: Device: Nicom (TM)

INTERVENTIONS:
Device: Nicom (TM) — Heart rate, arterial pressure and cardiac output measurements (monitor NICOM) performed in the dorsal decubitus position and in the left lateral decubitus

SUMMARY:
Fetal heart rate abnormalities are common. Miller et al. have demonstrated that new onset fetal heart rate abnormalities after initial labor epidural dosing occur more frequently in women with a low admission pulse pressure than those with a normal admission pulse. The aim of the present study is to look for a statistical link between the occurrence of a fetal heart abnormality requiring an intervention and maternal hemodynamic factors (blood pressure, pulse pressure, and cardiac output) measured before epidural analgesia in two positions: dorsal decubitus position and in the left lateral decubitus.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* gestational age ≥ 36 weeks
* single eutrophic fetus
* wishing for epidural analgesia
* cervical dilatation less than or equal to 5 cm
* spontaneous labor
* scheduled for a vaginal delivery.

Non-inclusion Criteria:

* prematurity (< 36 weeks of amenorrhea) or post-term birth
* intention of induction of labour using oxytocin before epidural analgesia or prostaglandin
* contraindication to epidural analgesia
* history of hypertension or gravidic hypertension or heart disorder
* gestational diabetes
* foetal malformation or oligohydramnios or fetal growth abnormality
* fœtal macrosomia diagnosed by ultrasonic scanning
* hematocrit less than 20%

Exclusion Criteria

* induction of labour using oxytocin before epidural analgesia
* newborn weight > 4kg at birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Fetal heart rate | 4 days
  Fetal heart rate abnormalities occurring during the first hour of epidural analgesia and requiring an intervention. Relationship between maternal hemodynamic factors (heart rate, blood pressure, pulse pressure, and cardiac output) measured before epidural analgesia in two positions (dorsal decubitus position and in the left lateral decubitus) and fetal heart rate abnormalities occurring during the first hour of epidural analgesia and requiring an intervention.

SECONDARY OUTCOMES:
Fetal heart rate | 4 days
  Fetal heart rate abnormalities occurring during the labor (>1 hour) and requiring an intervention. Comparison of the prognostic performance of pulse pressure and cardiac output to detect fetal heart rate abnormalities
Mode of delivery | 4 days
  Relationship between maternal hemodynamic factors (heart rate, blood pressure, pulse pressure, and cardiac output) measured before epidural analgesia in two positions (dorsal decubitus position and in the left lateral decubitus) and mode of delivery.
Newborn heart rate, blood pressure, pulse pressure, and cardiac output | 4 days
  Relationship between maternal hemodynamic factors (heart rate, blood pressure, pulse pressure, and cardiac output) measured before epidural analgesia in two positions (dorsal decubitus position and in the left lateral decubitus) and newborn health status.
Number of patients with hemodynamic abnormalities | 4 days
  Heart rate, blood pressure, pulse pressure, and cardiac output measured before and after epidural analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Le Guen, MD, Principal Investigator — Hôpital Foch; Marc Fischler, MD PhD, Study Chair — Hôpital Foch; Frédéric Mercier, MD PhD, Study Chair — AP-HP Hôpital A. Béclère
Locations (4):
- France (4):
  - AP-HP Hopital Antoine Beclere, Clamart
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Institut Mutualiste Montsouris, Paris
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller NR, Cypher RL, Nielsen PE, Foglia LM. Maternal pulse pressure at admission is a risk factor for fetal heart rate changes after initial dosing of a labor epidural: a retrospective cohort study. Am J Obstet Gynecol. 2013 Oct;209(4):382.e1-8. doi: 10.1016/j.ajog.2013.05.049. Epub 2013 Jun 13. PMID 23769849